CLINICAL TRIAL: NCT03736161
Title: Safety and Efficacy of Tofacitinib vs Methotrexate in the Treatment of Psoriatic Arthritis
Acronym: PsOLSET-BD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Globe Pharmaceuticals Limited (Other)
Responsible Party: Principal Investigator, Dr. Prayush Sharma, Principal investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PsOLSET-BD
Record Dates: First submitted 2018-11-02; First posted 2018-11-09 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Psoriatic Arthritis
Keywords: PsA
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — tofacitinib; Methotrexate

STUDY DESIGN:
Intervention Model Description: Open label randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A- Tofacitinib (Experimental): Tofacitinib 5mg twice daily orally. Patients with inadequate response to Tofacitinib 5 mg BD at the end of 3 months will be put on Tofacitinib 10 mg BD.
  Interventions: Drug: Group A- Tofacitinib
- Group B- Methotrexate (Placebo Comparator): Methotrexate in increasing dose starting from 15 mg weekly to a maximum dose of 25 mg weekly from the end of 1st month. Patients with inadequate response to highest dose of MTX at the end of 3 months will be put on Tofacitinib 5 mg BD.
  Interventions: Drug: Group B- Methotrexate

INTERVENTIONS:
Drug: Group A- Tofacitinib — Group A patients will receive Tofacitinib 5mg BD. Patients will be followed up at 1, 3 and 6 months. Patients with inadequate response to Tofacitinib 5 mg BD at the end of 3 months will be put on Tofacitinib 10 mg BD. Primary endpoint for efficacy will be determined by ACR 20 response.
  Other Names: Tofacitinib
  Arms: Group A- Tofacitinib
Drug: Group B- Methotrexate — Group B patients will receive Methotrexate in increasing dose weekly with maximum dose up to 25 mg/week. Patients will be followed up at 1, 3 and 6 months. Patients with inadequate response to highest dose of MTX at the end of 3 months will be put on Tofacitinib 5 mg BD. Primary endpoint for efficacy will be determined by ACR 20 response.
  Other Names: Methotrexate
  Arms: Group B- Methotrexate

SUMMARY:
Title Safety and Efficacy of Tofacitinib vs Methotrexate in the treatment of Psoriatic Arthritis- An Open Label Randomized single center study Psoriatic arthritis is defined as an inflammatory arthropathy associated with skin psoriasis and usually negative for rheumatoid factor. Till date, many NSAIDs, corticosteroids, DMARDs have been used, but the safety and efficacy issues demands more researches. The prevalence of PsA worldwide is about 1%-2% and among patients with psoriasis ranges from 7% to 42%. The pathogenesis of PsA involves many cytokines. Tofacitinib is an oral Janus Kinase (JAK) inhibitor with immunomodulatory and anti-inflammatory mechanism. It binds to JAK and prevents the activation of the JAK-signal transducers and activators of transcription (STAT) signaling pathway which ultimately decreases the production of pro-inflammatory cytokines, and prevents both inflammatory response and the inflammation-induced damage. It has shown better efficacy in many diseases like Rheumatoid Arthritis, Axial spondyloarthropathies, Psoriasis, Psoriatic Arthritis, Alopecia areata, dry eye disease.

This prospective, open label, randomized study will be conducted in inpatient and outpatient departments of Rheumatology, BSMMU, Dhaka, Bangladesh in 110 adult volunteers (>18 years) of both genders diagnosed as psoriatic arthritis. Patients will be divided equally into two groups, Group A will be put on Tofacitinib 5 mg twice daily and Group B will be put on Methotrexate weekly in increasing dose with maximum dose of 25 mg weekly. Groups will be divided on the basis of randomization by random number table. Patients with inadequate response to highest dose of MTX or Tofacitinib 5 mg BD at the end of 3 months will be put on Tofacitinib 5 mg BD or Tofacitinib 10 mg BD respectively. The patients not eligible for therapy will not be included in the study. Patients will be followed up at 1, 3 and 6 months. Baseline characteristics will be monitored and recorded at 3 and 6 months.

The clinical information of the study subjects will be recorded in a structured history, clinical examination and questionnaire. All subjects will be enrolled after having informed written consent. The participants will enjoy every right to participate or withdraw from the study at any point of time. Response to Tofacitinib will be expressed in mean, standard deviation and percentage. Ethical clearance will be taken from the Institutional Review Board (IRB) of BSMMU.

DETAILED DESCRIPTION:
Background:

Methotrexate, an anti-folate drug, is a widely accepted and commonly used DMARD for the treatment of PsA. Tofacitinib is a JAK inhibitor, and relatively new drug for this condition.

Aims:

To assess and compare safety and efficacy of Tofacitinib and Methotrexate in the treatment of PsA.

Methodology:

This open label, randomized, prospective study was conducted in Department of Rheumatology, BSMMU, Dhaka for 1½ years from September, 2017 to February, 2019. 61 patients, aged >18 years with the diagnosis of PsA for ≥3 months were randomized into two groups. 29 patients (Tofacitinib 5mg BD) and 32 patients (MTX from 15 mg/week to 25 mg/week over 1 month) were enrolled and followed-up at the end of 1, 3 and 6 months. Primary endpoint was ACR 20 response at the end of 3 months. Patients who achieved treatment target on the basis of DAPSA score at the end of 3 months were allowed to continue previuos treatment and assessed for safety and efficacy till 6 months. Patients not achieving treatment target in Tofacitinib group were put on Tofacitinib 10 mg BD and in MTX group were put on Tofacitinib 5 mg BD. These patients were followed-up for safety and efficacy at the end of 6 months. Secondary outcome measures were EULAR response, 66/68 joints SJC/TJC, VAS for pain, ESR, CRP, DAPSA, DAS28, PASI, PASI 75 response, MASES and HAQ-DI. Safety assessment was done on the basis of clinical history, examination and laboratory findings at each follow-up. Ethical clearance was obtained from IRB, BSMMU at the beginning. Statistical analysis was done using chi-square test, Fisher's exact test, paired sample t-test and independent sample t-test. Missing data were dealt with intention to treat (ITT) analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients more than 18 years
2. Psoriatic arthritis > 3 months with peripheral involvement diagnosed on the basis of CASPAR criteria
3. Unresponsive to more than 2 NSAIDs at maximum recommended doses for more than 4 weeks, i.e 2 weeks for each NASID

5. Patients with active disease 6. PsA with or without extra-articular features like enthesitis, dactylitis and nail changes

Exclusion Criteria:

1. Systemic infections requiring hospital admission during the past 6 months
2. A history of active infectious disorders (including active or latent tuberculosis), and/or a history of chronic or recurrent serious infective diseases, opportunistic infections
3. Hemoglobin (Hb) < 9 g/dl
4. White blood cell count < 3000, Neutrophil count < 1000, Platelet count < 100000
5. Live vaccines within 3 months prior to the first dose
6. Serum creatinine > upper limit of normal reference range
7. GFR less than 50 mL/min
8. Alanine aminotransaminase (ALT) more than 2 times of ULN
9. Pregnant or breast feeding, females of child-bearing potential not using highly effective contraception
10. New York Heart Association Class III and IV congestive heart failure
11. Evidence or history of malignancy, with the exception of adequately treated or excised non-metastatic basal or squamous cell cancer of the skin or cervical carcinoma in situ
12. Any lymphoproliferative disorder, history of lymphoma, leukemia, or signs and symptoms suggestive of current lymphatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-09-28 (Actual); Study Completion 2019-09-28 (Actual)

PRIMARY OUTCOMES:
American college of Rheumatology 20 (ACR 20) response | 3 months
  This response criteria is achieved if there is 20% improvement in tender or swollen joint counts along with 20% improvement in three of the following five parameters:
  1. Erythrocyte sedimentation rate in mm in 1st hour
  2. Patient assessment in numerical scale of 10 (range: 0-10)
  3. Physician assessment in numerical scale of 10 (range: 0-10)
  4. Visual analog pain scale (range: 0-10)
  5. Disability/functional questionnaire with maximum score of 3 (range: 0-3)

SECONDARY OUTCOMES:
Disease activity score-28 joint-ESR score (DAS28-ESR) | 1, 3 and 6 months
  Disease activity score for assessment of disease activity of rheumatoid arthritis. It is calculated using the following parameters:
  1. Tender joint count- 28 joints
  2. Swollen joint count- 28 joints
  3. Patient global assessment (range 1-10)
  4. Erythrocyte sedimentation rate in mm in 1st hour Greater score means poor prognosis.A score of greater than 5.1 implies active disease, less than 3.2 low disease activity, and less than 2.6 remission.
Disease activity index for psoriatic Arthritis (DAPSA) | 1, 3 and 6 months
  The DAPSA score consists of five variables: tender and swollen joints (TJC68, SJC66), patient global assessment and patient pain assessment (each on a 10-cm visual analogue scale [VAS]), and CRP. The addition of these variables is the result.
  Disease Activity: 0-4 Remission, 5-14 low, 15-28 moderate, >28 high Disease Activity
Psoriasis Area and Severity Index (PASI) | 1, 3 and 6 months
  PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease).
  The body is divided into four sections (head (H) (10% of a person's skin); arms (A) (20%); trunk (T) (30%); legs (L) (40%)). Each of these areas is scored by itself, and then the four scores are combined into the final PASI. For each section, the percent of area of skin involved, is estimated and then transformed into a grade from 0 to 6:
  1. 0% of involved area
  2. < 10% of involved area
  3. 10-29% of involved area
  4. 30-49% of involved area
  5. 50-69% of involved area
  6. 70-89% of involved area
  7. 90-100% of involved area Within each area, the severity is estimated by three clinical signs: erythema, induration and desquamation.
Maastricht Ankylosing Spondylitis Enthesitis Score | 1, 3 and 6 months
  The Maastricht Ankylosing Spondylitis Enthesitis Score uses 13 most speciﬁc and sensitive sites. These include the bilateral ﬁrst and seventh costochondral joints, the anterior and posterior superior iliac spines, the iliac crests, the ﬁfth lumbar spinous process, and the proximal insertion of Achilles tendon.
  Total score-13 Range: 0-13 Greater score implies greeater entheses involvement, and thus greater disease activity.
Health Assessment Questionnaire- Disability Index | 1, 3 and 6 months
  An assessment tool for chronic diseases. A questionnaire where a person indicates the amount of difficulty they have with: dressing and grooming, arising, eating, walking, hygiene, reaching, gripping and performing common daily activities.
  Total score- 3 Range- 0-3 Higher scores indicates higher disability.
EULAR response | 3 months
  EULAR response according to predefined changes in DAS28-ESR scores
66/68 joints SJC/TJC | 1, 3 and 6 months
  SJC- swollen joint count and TJC- tender joint count
ESR | 1, 3 and 6 months
  Erythrocyte sedimentation rate
CRP | 1, 3 and 6 months
  C-reactive protein
PASI75 response | 3 and 6 months
  75% improvement in PASI score

CONTACTS AND LOCATIONS:
Overall Officials: Prayush Sharma, MD, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jandus C, Bioley G, Rivals JP, Dudler J, Speiser D, Romero P. Increased numbers of circulating polyfunctional Th17 memory cells in patients with seronegative spondylarthritides. Arthritis Rheum. 2008 Aug;58(8):2307-17. doi: 10.1002/art.23655. PMID 18668556
- [Background] Ghoreschi K, Jesson MI, Li X, Lee JL, Ghosh S, Alsup JW, Warner JD, Tanaka M, Steward-Tharp SM, Gadina M, Thomas CJ, Minnerly JC, Storer CE, LaBranche TP, Radi ZA, Dowty ME, Head RD, Meyer DM, Kishore N, O'Shea JJ. Modulation of innate and adaptive immune responses by tofacitinib (CP-690,550). J Immunol. 2011 Apr 1;186(7):4234-43. doi: 10.4049/jimmunol.1003668. Epub 2011 Mar 7. PMID 21383241
- [Background] Moll JM, Wright V. Familial occurrence of psoriatic arthritis. Ann Rheum Dis. 1973 May;32(3):181-201. doi: 10.1136/ard.32.3.181. No abstract available. PMID 4715537
- [Background] Ritchlin C, Haas-Smith SA, Hicks D, Cappuccio J, Osterland CK, Looney RJ. Patterns of cytokine production in psoriatic synovium. J Rheumatol. 1998 Aug;25(8):1544-52. PMID 9712099
- [Background] Rosengren S, Corr M, Firestein GS, Boyle DL. The JAK inhibitor CP-690,550 (tofacitinib) inhibits TNF-induced chemokine expression in fibroblast-like synoviocytes: autocrine role of type I interferon. Ann Rheum Dis. 2012 Mar;71(3):440-7. doi: 10.1136/ard.2011.150284. Epub 2011 Nov 25. PMID 22121136
- [Background] Taylor W, Gladman D, Helliwell P, Marchesoni A, Mease P, Mielants H; CASPAR Study Group. Classification criteria for psoriatic arthritis: development of new criteria from a large international study. Arthritis Rheum. 2006 Aug;54(8):2665-73. doi: 10.1002/art.21972. PMID 16871531
- [Background] Langley RG, Krueger GG, Griffiths CE. Psoriasis: epidemiology, clinical features, and quality of life. Ann Rheum Dis. 2005 Mar;64 Suppl 2(Suppl 2):ii18-23; discussion ii24-5. doi: 10.1136/ard.2004.033217. PMID 15708928
- [Background] Gladman DD, Antoni C, Mease P, Clegg DO, Nash P. Psoriatic arthritis: epidemiology, clinical features, course, and outcome. Ann Rheum Dis. 2005 Mar;64 Suppl 2(Suppl 2):ii14-7. doi: 10.1136/ard.2004.032482. PMID 15708927
- [Background] Sherlock JP, Joyce-Shaikh B, Turner SP, Chao CC, Sathe M, Grein J, Gorman DM, Bowman EP, McClanahan TK, Yearley JH, Eberl G, Buckley CD, Kastelein RA, Pierce RH, Laface DM, Cua DJ. IL-23 induces spondyloarthropathy by acting on ROR-gammat+ CD3+CD4-CD8- entheseal resident T cells. Nat Med. 2012 Jul 1;18(7):1069-76. doi: 10.1038/nm.2817. PMID 22772566
- [Background] Partsch G, Steiner G, Leeb BF, Dunky A, Broll H, Smolen JS. Highly increased levels of tumor necrosis factor-alpha and other proinflammatory cytokines in psoriatic arthritis synovial fluid. J Rheumatol. 1997 Mar;24(3):518-23. PMID 9058659
- [Background] Gossec L, Smolen JS, Ramiro S, de Wit M, Cutolo M, Dougados M, Emery P, Landewe R, Oliver S, Aletaha D, Betteridge N, Braun J, Burmester G, Canete JD, Damjanov N, FitzGerald O, Haglund E, Helliwell P, Kvien TK, Lories R, Luger T, Maccarone M, Marzo-Ortega H, McGonagle D, McInnes IB, Olivieri I, Pavelka K, Schett G, Sieper J, van den Bosch F, Veale DJ, Wollenhaupt J, Zink A, van der Heijde D. European League Against Rheumatism (EULAR) recommendations for the management of psoriatic arthritis with pharmacological therapies: 2015 update. Ann Rheum Dis. 2016 Mar;75(3):499-510. doi: 10.1136/annrheumdis-2015-208337. Epub 2015 Dec 7. PMID 26644232
- [Background] Maeshima K, Yamaoka K, Kubo S, Nakano K, Iwata S, Saito K, Ohishi M, Miyahara H, Tanaka S, Ishii K, Yoshimatsu H, Tanaka Y. The JAK inhibitor tofacitinib regulates synovitis through inhibition of interferon-gamma and interleukin-17 production by human CD4+ T cells. Arthritis Rheum. 2012 Jun;64(6):1790-8. doi: 10.1002/art.34329. Epub 2011 Dec 6. PMID 22147632
- [Background] Kane D, Jensen LE, Grehan S, Whitehead AS, Bresnihan B, Fitzgerald O. Quantitation of metalloproteinase gene expression in rheumatoid and psoriatic arthritis synovial tissue distal and proximal to the cartilage-pannus junction. J Rheumatol. 2004 Jul;31(7):1274-80. PMID 15229943
- [Background] Smolen JS, Aletaha D, Gruben D, Zwillich SH, Krishnaswami S, Mebus C. Brief Report: Remission Rates With Tofacitinib Treatment in Rheumatoid Arthritis: A Comparison of Various Remission Criteria. Arthritis Rheumatol. 2017 Apr;69(4):728-734. doi: 10.1002/art.39996. Epub 2017 Mar 8. PMID 27907269
- [Background] Helliwell P, Coates LC, FitzGerald O, Nash P, Soriano ER, Elaine Husni M, Hsu MA, Kanik KS, Hendrikx T, Wu J, Kudlacz E. Disease-specific composite measures for psoriatic arthritis are highly responsive to a Janus kinase inhibitor treatment that targets multiple domains of disease. Arthritis Res Ther. 2018 Oct 29;20(1):242. doi: 10.1186/s13075-018-1739-0. PMID 30373651
- [Background] Olivieri I, Giasi V, Scarano E, Gigliotti P, D'Angelo S, Padula A. A brief course of anti-TNF-alpha therapy can cure recurrent episodes of HLA-B27-associated severe and refractory heel enthesitis. Clin Exp Rheumatol. 2009 Nov-Dec;27(6):1057; author reply 1058. No abstract available. PMID 20149333
- [Background] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Thirunavukkarasu K, DeMasi R, Geier J, Kwok K, Wang L, Riese R, Wollenhaupt J. Long-term safety of tofacitinib for the treatment of rheumatoid arthritis up to 8.5 years: integrated analysis of data from the global clinical trials. Ann Rheum Dis. 2017 Jul;76(7):1253-1262. doi: 10.1136/annrheumdis-2016-210457. Epub 2017 Jan 31. PMID 28143815
- [Result] Gladman DD, Shuckett R, Russell ML, Thorne JC, Schachter RK. Psoriatic arthritis (PSA)--an analysis of 220 patients. Q J Med. 1987 Feb;62(238):127-41. PMID 3659255
- [Result] Fraser AD, van Kuijk AW, Westhovens R, Karim Z, Wakefield R, Gerards AH, Landewe R, Steinfeld SD, Emery P, Dijkmans BA, Veale DJ. A randomised, double blind, placebo controlled, multicentre trial of combination therapy with methotrexate plus ciclosporin in patients with active psoriatic arthritis. Ann Rheum Dis. 2005 Jun;64(6):859-64. doi: 10.1136/ard.2004.024463. Epub 2004 Nov 4. PMID 15528283
- [Result] Coates LC, Helliwell PS. Methotrexate Efficacy in the Tight Control in Psoriatic Arthritis Study. J Rheumatol. 2016 Feb;43(2):356-61. doi: 10.3899/jrheum.150614. Epub 2015 Dec 15. PMID 26669913
- [Result] Mease P, Hall S, FitzGerald O, van der Heijde D, Merola JF, Avila-Zapata F, Cieslak D, Graham D, Wang C, Menon S, Hendrikx T, Kanik KS. Tofacitinib or Adalimumab versus Placebo for Psoriatic Arthritis. N Engl J Med. 2017 Oct 19;377(16):1537-1550. doi: 10.1056/NEJMoa1615975. PMID 29045212
- [Result] Gladman D, Rigby W, Azevedo VF, Behrens F, Blanco R, Kaszuba A, Kudlacz E, Wang C, Menon S, Hendrikx T, Kanik KS. Tofacitinib for Psoriatic Arthritis in Patients with an Inadequate Response to TNF Inhibitors. N Engl J Med. 2017 Oct 19;377(16):1525-1536. doi: 10.1056/NEJMoa1615977. PMID 29045207
- [Result] Baranauskaite A, Raffayova H, Kungurov NV, Kubanova A, Venalis A, Helmle L, Srinivasan S, Nasonov E, Vastesaeger N; RESPOND investigators. Infliximab plus methotrexate is superior to methotrexate alone in the treatment of psoriatic arthritis in methotrexate-naive patients: the RESPOND study. Ann Rheum Dis. 2012 Apr;71(4):541-8. doi: 10.1136/ard.2011.152223. Epub 2011 Oct 12. PMID 21994233
- [Result] Kingsley GH, Kowalczyk A, Taylor H, Ibrahim F, Packham JC, McHugh NJ, Mulherin DM, Kitas GD, Chakravarty K, Tom BD, O'Keeffe AG, Maddison PJ, Scott DL. A randomized placebo-controlled trial of methotrexate in psoriatic arthritis. Rheumatology (Oxford). 2012 Aug;51(8):1368-77. doi: 10.1093/rheumatology/kes001. Epub 2012 Feb 17. PMID 22344575
- [Result] Dalrymple JM, Stamp LK, O'Donnell JL, Chapman PT, Zhang M, Barclay ML. Pharmacokinetics of oral methotrexate in patients with rheumatoid arthritis. Arthritis Rheum. 2008 Nov;58(11):3299-308. doi: 10.1002/art.24034. PMID 18975321
- [Result] Fleischmann R, Wollenhaupt J, Takiya L, Maniccia A, Kwok K, Wang L, van Vollenhoven RF. Safety and maintenance of response for tofacitinib monotherapy and combination therapy in rheumatoid arthritis: an analysis of pooled data from open-label long-term extension studies. RMD Open. 2017 Dec 18;3(2):e000491. doi: 10.1136/rmdopen-2017-000491. eCollection 2017. PMID 29435359
- [Result] Van Vollenhoven, R.F., Wallenstein, G., Lee, E.B., Fleischmann, R., Zwillich, S.H., Gruben, D., Koncz, T., Bradley, J., Wilkinson, B. and Strand, V., 2013. THU0151 Effects of tofacitinib (CP-690,550), an oral janus kinase inhibitor, or adalimumab on patient reported outcomes in a phase 3 study of active rheumatoid arthritis. Annals of the Rheumatic Diseases, 71(Suppl 3), pp.206-206.
- [Result] Strober B, Teller C, Yamauchi P, Miller JL, Hooper M, Yang YC, Dann F. Effects of etanercept on C-reactive protein levels in psoriasis and psoriatic arthritis. Br J Dermatol. 2008 Aug;159(2):322-30. doi: 10.1111/j.1365-2133.2008.08628.x. Epub 2008 May 22. PMID 18503600
- [Result] Tsakok T, Jabbar-Lopez ZK, Smith CH. Subcutaneous methotrexate in patients with moderate-to-severe psoriasis: a critical appraisal. Br J Dermatol. 2018 Jul;179(1):50-53. doi: 10.1111/bjd.16424. Epub 2018 May 9. PMID 29399784
- [Result] Paul C, Cather J, Gooderham M, Poulin Y, Mrowietz U, Ferrandiz C, Crowley J, Hu C, Stevens RM, Shah K, Day RM, Girolomoni G, Gottlieb AB. Efficacy and safety of apremilast, an oral phosphodiesterase 4 inhibitor, in patients with moderate-to-severe plaque psoriasis over 52 weeks: a phase III, randomized controlled trial (ESTEEM 2). Br J Dermatol. 2015 Dec;173(6):1387-99. doi: 10.1111/bjd.14164. Epub 2015 Nov 7. PMID 26357944
- [Result] van der Heijde D, Deodhar A, Wei JC, Drescher E, Fleishaker D, Hendrikx T, Li D, Menon S, Kanik KS. Tofacitinib in patients with ankylosing spondylitis: a phase II, 16-week, randomised, placebo-controlled, dose-ranging study. Ann Rheum Dis. 2017 Aug;76(8):1340-1347. doi: 10.1136/annrheumdis-2016-210322. Epub 2017 Jan 27. PMID 28130206
- [Result] 31. McInnes IB, Mease PJ, Kirkham B, Kavanaugh A, Ritchlin CT, Rahman P, et al. Secukinumab, a human anti-interleukin-17A monoclonal antibody, improves active psoriatic arthritis: 24-week efficacy and safety data from a phase 3 randomized, multicenter, double-blind, placebo-controlled study using subcutaneous dosing [abstract]. Arthritis Rheumatol. 2014; 66:3529. 92.
- [Result] Kavanaugh A, Mease PJ, Gomez-Reino JJ, Adebajo AO, Wollenhaupt J, Gladman DD, Hochfeld M, Teng LL, Schett G, Lespessailles E, Hall S. Longterm (52-week) results of a phase III randomized, controlled trial of apremilast in patients with psoriatic arthritis. J Rheumatol. 2015 Mar;42(3):479-88. doi: 10.3899/jrheum.140647. Epub 2015 Jan 15. PMID 25593233
- [Result] Salliot C, van der Heijde D. Long-term safety of methotrexate monotherapy in patients with rheumatoid arthritis: a systematic literature research. Ann Rheum Dis. 2009 Jul;68(7):1100-4. doi: 10.1136/ard.2008.093690. Epub 2008 Dec 5. PMID 19060002
- See also: Safety, efficacy and tolerability of oral tofacitinib in Japanese patients with psoriasis and psoriatic arthritis — https://www.ncbi.nlm.nih.gov/pubmed?term=2016%5Bpdat%5D+AND+Asahina%2C+Akihiko%5Bauthor%5D+AND+Oral+tofacitinib+efficacy%2C+safety+and+tolerability&TransSchema=title&cmd=detailssearch
- See also: Modulation of innate and adaptive immune by Tofacitinib — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3108067/
- See also: EULAr 2015 recommendations for the treatment of Psoriatic Arthritis — https://ard.bmj.com/content/75/3/499
- See also: Pfizer's poster and oral presentation at ACR conference — https://www.pfizer.com/news/press-release/press-release-detail/pfizer_announces_results_from_phase_3_opal_clinical_development_program_investigating_xeljanz_tofacitinib_citrate_for_psoriatic_arthritis